CLINICAL TRIAL: NCT06992843
Title: A Multicenter, Prospective, Stepped Wedge Cluster Randomized Controlled Study on the Effect of Neuroprotection Bundles on the Improvement of Neurological Outcomes After Cardiopulmonary Resuscitation
Brief Title: Neuroprotection Bundles For Comatose Survivors Following Cardiac Arrest
Acronym: LAPTOPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, icuzhanglina, Professor, Xiangya Hospital of Central South University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 2024121757
Record Dates: First submitted 2025-05-06; First posted 2025-05-28 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-07

CONDITIONS: Cardiac Arrest; Post-cardiac Arrest Care
Keywords: post-cardiac arrest care; neuroprotection; cardiac arrest; Care Bundle; Clinical Trial; Stepped-wedge Cluster
MeSH Terms: conditions — Heart Arrest | interventions — Neuroprotection

STUDY DESIGN:
Intervention Model Description: Stepped-wedge Cluster Randomised Trial
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Goal-directed care bundle for neuroprotection (Other): Management policy to receive a goal-directed care bundle that involves the rapid correction (<24 hour) of physiological variables as soon as the abnormality is recognised and for the control to be maintained in patients for 72h or hospital discharge (or death, if sooner)
  Interventions: Other: Goal-directed care bundle for neuroprotection
- Usual care group (Other): Patients receive the usual management based on local guidelines and hospital's individual policy.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Goal-directed care bundle for neuroprotection — Reducing lactate (Lac) to <2 mmol/L within 24 hours.Maintaining systolic arterial pressure at 120-140 mmHg.
  Elevating the head-of-bed to 30 degrees. Maintaining body temperature ≤37.7°C. Maintaining PaO₂ at 70-100 mmHg. Maintaining PaCO₂ at 35-45 mmHg. Maintaining blood glucose at 7.8-10.0 mmol/L. Maintaining serum sodium level at 140-150 mmol/L. If any management parameter falls outside the target range, immediate correction is required within 24 hours of enrollment and must be sustained for 72 hours. Given the dynamic nature of some targets (e.g., mean arterial pressure, body temperature), a degree of flexibility is permitted in achieving these goals. Patients are considered to have successfully implemented the neuroprotection bundle if the achievement rate of individual targets is ≥80% and all targets are met. The medications(antipyretics, vasopressor agents) is acceptable to achieve these targets.
  Arms: Goal-directed care bundle for neuroprotection
Other: Usual Care — Usual care decisions about the location of care delivery, investigations, monitoring, and all treatments will be made by the treating clinical team.
  Arms: Usual care group

SUMMARY:
The investigators designed LAPTOPS to determine the effectiveness of a goal-directed neuroprotection bundles of active management including body temperature,PaCO2,PaO2,position,Blood glucose ,blood sodium,Blood pressure and Lactate vs. usual care in adult post-cardiac arrest care.

LAPTOPS is a large-scale pragmatic clinical trial to provide reliable evidence over the effectiveness of a widely applicable goal-directed care bundle in acute phase of adult post-cardiac arrest care.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and < 80 years
* Patients of in-hospital or out-of-hospital cardiac arrest who have returned -spontaneous circulation (ROSC) after cardiopulmonary resuscitation and do not require CPR for more than 20 minutes;
* Patients who are unconscious after ROSC, defined as FOUR motor response score < 4 points or GSC ≤ 8 points;
* Family members or legal representatives signed informed consent.

Exclusion Criteria:

* Unwitnessed cardiac arrest, estimated time from cardiac arrest to start of CPR > 30 minutes;
* Time from cardiac arrest to ROSC > 60 minutes;
* Patients who woke up immediately after ROSC by CPR;
* End-stage diseases;
* Cardiac arrest considered to be caused by neurological diseases;
* The patient was in a vegetative state before cardiac arrest;
* The interval from the onset of cardiac arrest to enrollment is >72 hours .

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1008 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Favorable neurological prognosis | 90 days post cardiac arrest
  Assessed using the CPC score, with a score of 1-2 being a favorable outcome.

SECONDARY OUTCOMES:
GCS score | 7 days post cardiac arrest
  GCS score
CPC score | 1 day (discharge date)
  CPC score
GCS score | 1 day (discharge date)
  GCS score
Time to death | 180 days
  Number of days alive within 180 days from ROSC.
the length of ICU stay | The total length of IC-stay will be determined from the date of ICU admission until the patient is discharged from the Intensive Care Unit or the date of death from any cause, assessed up to 1 year after the first day of admission.
  the length of ICU stay
the length of hospital stay | The total length of hospital-stay will be determined from the date of ICU admission until the patient is discharged from the hospital or the date of death from any cause assessed up to 1 year after the first day of admission.
  the length of hospital stay
the length of mechanical ventilation | Total ventilation time during ICU stay will be determined when the patient is discharged from the ICU or when the patient past away from any cause, assessed up to 1 year after the first day of admission.
  the length of mechanical ventilation
the incidence of adverse event | From the date of ICU admission until the patient is discharged from the Intensive Care Unit or the date of death from any cause, assessed up to 1 year after the first day of admission.
  The incidence of adverse effects during ICU treatment
in-hospital mortality | The total length of hospital-stay will be determined from the date of ICU admission until the patient is discharged from the hospital or the date of death from any cause assessed up to 1 year after the first day of admission.
  in-hospital mortality
28-day mortality | 28 days post cardiac arrest
  28-day mortality
Quality of life assessment | 90 days post cardiac arrest
  Health-related Quality of Life - EQ-5D (Index value)
bundle compliance rate | 72 hours
  referring to the proportion of patients whose management parameters are within the target ranges.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya hospital，Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No